CLINICAL TRIAL: NCT03244163
Title: Randomized Controlled Trial of Spyglass DS Peroral Cholangioscope Guided Laser Lithotripsy or Electrohydraulic Lithotripsy Versus Conventional Basket Mechanical Lithotripsy for Endoscopic Removal of Complicated Bile Duct Stones
Brief Title: Spyglass DS Peroral Cholangioscope Guided LL or EHL Versus BML for Endoscopic Removal of Complicated Bile Duct Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHOOT study
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Biliary Stones
Keywords: Spyglass DS; Laser lithotripsy; Endoscopic retrograde cholangiopancreatography
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LASER ARM (Experimental): Spyglass DS cholangioscope guided laser or electrohydraulic lithotripsy
  Interventions: Device: Spyglass DS cholangioscope
- CONVENTIONAL ARM (Active Comparator): Stone removal by conventional techniques, for example BML, without laser lithotripsy
  Interventions: Device: BML

INTERVENTIONS:
Device: Spyglass DS cholangioscope — The 1.8Fr holmium:YAG laser fiber (Lumenis, Yokneam, Israel) will be inserted into the cholangioscope's working channel for lithotripsy under direct visualization. An EHL probe may alternatively be used depending on availability. Lithotripsy is applied until fragments of the targeted stone are no longer lumen filling, and can be dispersed easily with fluid irrigation. Fragmented stones are then removed by a combination of conventional techniques. To confirm stone clearance, the Spyglass DS cholangioscope will be re-introduced, and the bile duct will be examined for residual stones from the confluence of the right and left intrahepatic ducts to the papillary opening
  Arms: LASER ARM
Device: BML — Biliary sphincterotomy with/without EPBD to the size of the lower bile duct with a limit of 15mm will be performed. Stones are removed by a combination of conventional BML, extraction balloon and/or baskets, without laser lithotripsy. An occlusion cholangiogram is performed to confirm stone clearance. In cases where stone clearance is incomplete, a plastic biliary stent bridging the stone will be inserted for temporary drainage until definitive management, usually within one month.
  Arms: CONVENTIONAL ARM

SUMMARY:
This study aims to compare the overall rate of endoscopic clearance of complicated bile duct stones by Spyglass DS peroral cholangioscopy guided holmium:YAG laser/electrohydraulic lithotripsy versus conventional BML.

DETAILED DESCRIPTION:
Currently, complicated bile duct stones are removed during endoscopic retrograde cholangiopancreatography (ERCP) by conventional mechanical lithotripsy, which means using a metal wire basket to capture the stone and crush it to make it easier to remove. This is successful in approximately 70% of patients, with the success rate inversely correlated to the size of the stone. Unsuccessful stone removal would require additional endoscopic, percutaneous or surgical interventions. Spyglass DS peroral cholangioscope-guided holmium:YAG laser/electrohydraulic lithotripsy is a recent alternate method for managing complicated bile duct stones. Also performed during ERCP, a thin flexible camera (called Spyglass DS peroral cholangioscope) is inserted into the bile duct to visualize the stone which can then be targeted by a laser beam for fragmentation (also known as laser lithotripsy). The smaller pieces are then removed. Direct comparisons of these procedures' efficacy however have not been performed.

The purpose of this study is to compare the efficacy and safety of Spyglass DS peroral cholangioscope-guided holmium:YAG laser/electrohydraulic lithotripsy (the laser arm) versus conventional basket mechanical lithotripsy alone (the conventional arm) for fragmentation and clearance of complicated bile duct stones.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complicated biliary stones
* Patients older than 18 years old
* Patients where informed consent can be obtained

Exclusion Criteria:

* Patients who cannot give informed consent
* Patients under 18 years old
* Pregnant or lactating patients
* Patient with altered gastrointestinal/biliary anatomy
* Patients with distal CBD malignant stricture from intrinsic or extrinsic causes
* Patients with ongoing cholangitis or biliary pancreatitis
* Patient with refractory bleeding tendencies (Platelet count <50,000/mm3 or International Normalized Ratio >1.5 despite correction with platelet or fresh frozen plasma transfusions)
* Patients with intrahepatic segmental stones
* Patients with contraindications to endoscopy due to comorbidities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-06-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall rate of endoscopic bile duct stone clearance | Intraoperative
  Overall rate of endoscopic bile duct stone clearance

SECONDARY OUTCOMES:
Technical feasibility | Intraoperative
  Technical feasibility defined as successful introduction of cholangioscope into the CBD, visualisation and laser targeting of stone
Incidence of adverse events | 30 days
  Incidence of adverse events
Need for and number of additional procedures for stone clearance | 6 months
  Need for and number of additional procedures for stone clearance

CONTACTS AND LOCATIONS:
Overall Officials: James LAU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: No